CLINICAL TRIAL: NCT07161661
Title: Feasibility of Implementing Manual Medicine in the Multimodal Management of Veterans and Service Members With Chronic Low Back Pain
Brief Title: Chronic Low Back Pain and Osteopathic Manipulation Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Clarence Nicodemus, VA WOC, Edward Hines Jr. VA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1850064-1; Department of Defense (Other Grant/Funding Number: CP230185)
Record Dates: First submitted 2025-09-02; First posted 2025-09-08 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Low Back Pain (CLBP); Low Back Pain
Keywords: Osteopathic manipulative treatment; Physical Medicine and Rehabilitation; Veterans; Osteopathic manipulation
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual VA Care Group (Active Comparator): All study participants will receive usual VA care that will be provided by a physiatrist at the Hines VA. After taking their medical history, they will perform a physical exam to assess their conditions. Based on the physical exam, the physicians may recommend more testing and/or treatment procedures.
  Interventions: Procedure: Usual VA Care
- Usual VA Care + OMT Group (Experimental): Participants in this group will receive your usual VA care plus OMT. The addition of OMT is the research portion of the treatment. During the physician prescribed usual care visits, participants will receive the OMT treatment. During OMT (the research portion), a physician may move participants muscles and joints using hands-on techniques including stretching, gentle pressure and resistance, as well as applying forces to specific areas of the body. While receiving OMT, participants may be asked to change positions such as standing, sitting, or lying on your back, stomach or side. This treatment will be provided by the VA physicians involved in this study.
  Interventions: Procedure: Usual VA Care; Procedure: Osteopathic manipulative treatment

INTERVENTIONS:
Procedure: Usual VA Care — The usual treatment provided by PM&R clinicians for CLBP
Procedure: Osteopathic manipulative treatment — Between your first visit (baseline) and 12 weeks, participants will receive up to 4 usual care visits plus OMT.
  Other Names: Osteopathic Neuromuscular Manipulative Medicine
  Arms: Usual VA Care + OMT Group

SUMMARY:
The goal of this clinical trial is to learn if adding Osteopathic Manipulative Therapy (OMT) to the usual medical care provided at the VA (usual VA care) improves treatment outcomes in individuals with chronic low back pain (CLBP). OMT is a set of hands-on techniques a doctor uses to move a patient's muscles and joints which include stretching, gentle pressure, resistance and applying forces to specific areas of the body. This feasibility clinical trial aims to learn about the treatment effects (e.g., effect sizes) of adding OMT to the usual medical care provided at the VA (Usual VA Care) in individuals with LBP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Seeking care for LBP from a participating VA clinic
* Able to follow study protocol
* Willing to be randomized to Usual VA Care or Usual VA Care + OMT
* Individuals with pain primarily in the LBP region lasting > 3 months and present on at least half the days during the past 6 months
* Pain rating over the past 7 days equal to or greater than 3/10 as indicated on the Numeric Rating Scale for Pain

Exclusion Criteria:

* Signs of serious pathology as a cause of LBP
* Underlying systemic or inflammatory conditions
* Neurological diseases
* Pregnancy
* Previous back surgery or spinal fracture within the past year
* Active workers' compensation or litigation for back pain
* Any conditions impeding study protocol implementation or contraindication to OMT
* No PM&R, OMT, chiropractic, or physical treatment where manual techniques are utilized within last 3mo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Low-Back Pain Specific Pain Intensity | Baseline, 12 weeks, and 24 weeks
  A numeric pain rating scale (NPRS) question adapted by the BACPAC to obtain pain rating for over last 7 days.

SECONDARY OUTCOMES:
Pain, Enjoyment, General Activity Scale (PEG) | Baseline, 12 weeks, and 24 weeks
  A 3-item measure to assess and to monitor different aspects of chronic pain. Originally intended to be used in a primary care setting, this instrument has been used as an outcome measure and recommended by NIH HEAL core outcome set.
Brief Pain Inventory (BPI) | Baseline, 12 weeks, and 24 weeks
  A 32-item questionnaire to assess pain history, interference, pain relief, pain quality, and perceived cause of pain.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, 12 weeks, and 24 weeks
  PROMIS Depression Short Form 4a (4 item) , PROMIS Short Form Anxiety 4a (4 item), PROMIS Physical Functioning 6b (6 item), PROMIS Sleep Disturbance 6a (6 item), PROMIS Fatigue 4a (4 item)
Patient Health Questionnaire (PHQ-2) | Baseline, 12 weeks, and 24 weeks
  2-item questionnaire to screen for depression symptoms (frequency of depressed mood and anhedonia) during the past 2 weeks.
Generalized Anxiety Disorder 2-item (GAD-2) | Baseline, 12 weeks, and 24 weeks
  A 2-item questionnaire to screen for generalized anxiety disorder, panic disorder, social anxiety disorder, and post-traumatic stress disorder.
Pain Catastrophizing Scale - Short Form 6 (PCS-6) | Baseline, 12 weeks, and 24 weeks
  A 6-item measure to assess catastrophizing of pain.
Sleep Duration | Baseline, 12 weeks, and 24 weeks
  A measure of duration to quantify the amount of sleep participants report, which is in addition to PROMIS Sleep Disturbance 6a.
Healthcare utilization cost | Baseline, 12 weeks, and 24 weeks
  The number of treatment visits and medication use during study enrollment
Patients' Global Impression of Change (PGIC) | Baseline, 12 weeks, and 24 weeks
  A 1-item questionnaire that measures perception of patients beliefs about the effectiveness of treatment.
Radicular Pain Questions | Baseline, 12 weeks, and 24 weeks
  A 2-item measure adapted from NIH Research Task Force to capture radicular symptoms below the knee and/or thigh.
Abbreviated Pain Somatization | Baseline, 12 weeks, and 24 weeks
  A 2-item measure that captures somatization of back pain as stomach pain and headaches.
Widespread Pain Inventory | Baseline, 12 weeks, and 24 weeks
  A 1-item question to document areas of pain other than the low back.
Low Back Pain Duration and Frequency | Baseline, 12 weeks, and 24 weeks
  A 2-item measure to document CLBP as defined by NIH Task Force (back pain lasting greater than or equal to 3 months and having LBP at least half the days in the past 6 months).
The Tobacco, Alcohol, Prescription medications, and other Substance Part 1 (TAPS1) | Baseline, 12 weeks, and 24 weeks
  A 5- item questionnaire to identify unhealthy substance.
Alcohol Use Disorders Identification Test (AUDIT-C) | Baseline, 12 weeks, and 24 weeks
  A 3-item alcohol screen that can help identify persons who are hazardous drinkers or have active alcohol use disorders.
Healing Encounters and Attitudes Lists (HEAL) | Baseline, 12 weeks, and 24 weeks
  A 39-item questionnaire to capture Patient-Provider Connection, Healthcare Environment, Treatment Expectancy, Positive Outlook, Spirituality, and Attitudes toward Complementary and Alternative Medicine (CAM)/CIH approaches.

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Hines, Jr. VA Hospital, PM&R Clinic, Hines, Illinois, United States